CLINICAL TRIAL: NCT00707850
Title: A Study on PEGASYS® (Peginterferon Alfa-2a (40KD)) Plus COPEGUS® (Ribavirin) in Iranian Thalassemic Patients With Chronic Hepatitis C Infection
Brief Title: Pegasys® Plus Ribavirin in Thalassemic Patients With Hepatitis C Virus Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Baqiyatallah Research Center for Gastroenterology and Liver Diseases (Other); Tehran Hepatitis Center (Other); Guilan University of Medical Sciences (Other); Tabriz Research Center for Gastroenterology and Liver Diseases (Unknown)
Responsible Party: Professor Seyed-Moayed Alavian, Baqiyatallah Research Center for Gastroenterology and Liver Diseases
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRCGL-08-06
Record Dates: First submitted 2008-06-26; First posted 2008-07-01 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2009-09

CONDITIONS: Hepatitis C; Thalassemia
Keywords: Hepatitis C; Thalassemia; Pegasys; Ribavirin
MeSH Terms: conditions — Hepatitis C; Thalassemia | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Thalassemic Patients with HCV
  Interventions: Drug: PEGASYS® (Peginterferon Alfa-2a (40KD)) Plus COPEGUS® (Ribavirin)

INTERVENTIONS:
Drug: PEGASYS® (Peginterferon Alfa-2a (40KD)) Plus COPEGUS® (Ribavirin) — PEGASYS: 180 microgram per week (Injection) Plus Ribavirin: [=<75 kg: 1000 mg; >75 kg: 1200 mg per day (PO)]
  Other Names: Peginterferon Alfa-2a (40KD) plus COPEGUS

SUMMARY:
Antiviral treatment of HCV in thalassemia has raised concerns of ribavirin-induced hemolysis and increased iron loading. Blood Transfusion in Thalassemic patients are a known high risk for acquiring hepatitis C. The investigators are trying the PEGASYS (Peginterferon alpha-2a(40 KD)) plus Ribavirin in Thalassemic patients with HCV.

DETAILED DESCRIPTION:
Patients with Thalassemia receive chronic blood transfusions and have an increased prevalence of chronic Hepatitis C virus (HCV) infection, particularly if transfused before HCV serological testing became available. The investigators enrolled 300 patients into the study. The patients received PEGASYS (Peginterferon alpha-2a(40 KD)) 180 microgram per week plus COPEGUS (Ribavirin) 1000 milligram for weight less than or equal 75 kg and 1200 milligram for more than 75 kg for 48 weeks. Follow up period is 6 months after treatment. The patients are visited every 4 weeks with biochemistry lab tests. The patients are checked with quantitative HCV RNA (Ribonucleic Acid) on the third months after initiation of the treatment to assess early virologic response and at the end of the study for complete response rate and on the six month after treatment completion for sustained response rate. The patients with undetectable HCV RNA are considered as responders.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA positive
* Age older than 12 years

Exclusion Criteria:

* Ongoing pregnancy or breast feeding
* History (Hx) of Hepatocellular Carcinoma (HCC)
* Hx of alcoholic liver disease
* Hx of bleeding from esophageal varices
* Hx of hemochromatosis
* Hx of autoimmune hepatitis
* Hx of Suicidal attempt
* Hx of cerebrovascular dis
* Hx of severe retinopathy
* Hx of severe psoriasis
* Hx of scleroderma
* Hx of metabolic liver disease
* Hx of Systemic Lupus Erythematosus (SLE)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Early Virologic Response | After 12 weeks of Treatment
End of Treatment Response | 48 Weeks
Sustained Virologic Response | 24 weeks after Treatment
Rapid Virologic Response | One month after Treatment

SECONDARY OUTCOMES:
Tolerability of drugs for whole therapy period | During Treatment
Biochemical response (ALT) | End of Treatment AND 24 weeks after Treatment
Laboratory Parameters | During Treatment AND End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seyed-Moayed Alavian, Professor, Study Chair — Baqiyatallah Research Center for Gastroenterology and Liver Disea; Seyyed Mohammad Miri, M.D., Study Director — Baqiyatallah Research Center for Gastroenterology and Liver Disea; Pegah Karimi, M.D., Principal Investigator — Baqiyatallah Research Center for Gastroenterology and Liver Diseases; Maryam Keshvari, M.D., Principal Investigator — Iranian blood Transfusion Research Center; Bita Behnava, M.D., Principal Investigator — Baqiyatallah Research Center for Gastroenterology and Liver Diseases; Mohammad Hossein Somi, M.D., Principal Investigator — Research Center for Gastroenterology and Hepatology, Tabriz University of Medical Sciences, Tabriz; Fariborz Mansour-Ghanaei, M.D., Principal Investigator — Gastroenterology and Liver Diseases, Gastrointestinal and Liver Diseases Research Center (GLDRC), Guilan University of Medical Sciences, Rasht, Iran
Locations (1):
- Baqiyatallah Research Center for Gastroenterology and Liver Diseases, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Harmatz P, Jonas MM, Kwiatkowski JL, Wright EC, Fischer R, Vichinsky E, Giardina PJ, Neufeld EJ, Porter J, Olivieri N; Thalassemia Clinical Research Network. Safety and efficacy of pegylated interferon alpha-2a and ribavirin for the treatment of hepatitis C in patients with thalassemia. Haematologica. 2008 Aug;93(8):1247-51. doi: 10.3324/haematol.12352. Epub 2008 Jun 12. PMID 18556414